CLINICAL TRIAL: NCT04469582
Title: The Association of Bullous Pemphigoid With Dipeptidyl-peptidase 4 Inhibitors: Α Ten-year Prospective Observational Study.
Brief Title: The Association of Bullous Pemphigoid With Dipeptidyl-peptidase 4 Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Associate professsor of Cardiology, University of Athens
Other Study IDs: BP-DPP4is
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conducted a prospective study which included all patients diagnosed with biopsy-proven BP in the Dermatology Department of Attikon hospital between April 1, 2009 and December 31, 2019. 113 consecutive patients with BP were identified. The investigators included the patients with type 2 diabetes and investigated the percentage of patients who were under treatment with DPP4-is. The specific DPP4-i prescribed was also documented.Medical information including patients' age, sex, other comorbidities and concomitant medications were also recorded. Furthermore, the investigators evaluated the effect of different types of treatment (topical steroids, systemic corticosteroids, immunosuppressive agents) on bullous pemphigoid.

DETAILED DESCRIPTION:
Bullous pemphigoid (BP) is the most common chronic autoimmune skin disease which is characterized by the presentation of subepidermical blisters and mostly affects elderly patients . Recent studies have suggested that dipeptidyl peptidase-4 inhibitors (DPP-4is), an incretin-based drug for type 2 diabetes, as possible predisposing agents of BP . The objective of the study was to estimate the association between the use of DPP-4is and the development of BP in the setting of a tertiary university hospital and to raise awareness for everyday clinical practice, both among dermatologists as well as all physicians following patients with diabetes The study was designed as an observational prospective study.In the study included all patients who received a new diagnosis of BP and hospitalized in the Dermatology Department of our hospital between April 1, 2009 and December 31, 2019 Inclusion Criteria included a) biopsy proven bullous pemphigoid b) severe bullous pemphigoid c) recent manifestation of bullous pemphigoid (last four months).Exclusion Criteria included a) non bullous pemphigoid b) presentation of bullous pemphigoid more than four months c) treatment with DPP4is more than two years.

Overall, 113 consecutive patients with the diagnosis of BP were enrolled in the study.The investigators reviewed the percentage of patients with type 2 diabetes among all patients with BP.The number of patients who were under treatment with DPP4-is and the specific type of DPP4-is prescribed were also examined.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven bullous pemphigoid
* severe bullous pemphigoid
* recent manifestation of bullous pemphigoid (last four months)

Exclusion Criteria:

* non bullous pemphigoid
* presentation of bullous pemphigoid more than four months
* treatment with DPP4is more than two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the study included all patients diagnosed with biopsy-proven BP in the Dermatology Department of Attikon hospital between April 1, 2009 and December 31, 2019.
Sampling Method: Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2009-04-01 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Τhe correlation between the use of DPP-4is and the development of Bullous pemphigoid | baseline
  The investigators assessed the percentage of patients who were under treatment with DPP4-is among patients with bullous pemphigoid

CONTACTS AND LOCATIONS:
Overall Officials: Vaia Lambadiari, MD,PhD, Principal Investigator — 2nd department of internal medicine,University of Athens,Greece; Evangelia Papadavid, MD,PhD, Principal Investigator — 2nd department of dermatology and venereology,University of Athens, Greece; Aikaterini Kountouri, MD, Principal Investigator — 2nd department of internal medicine,University of Athens,Greece; Emmanouil Korakas, MD, Principal Investigator — 2nd department of internal medicine,University of Athens,Greece; Sofia Theotokoglou, Principal Investigator — 2nd department of dermatology and venereology,University of Athens, Greece; Konstantinos Theodoropoulos, Principal Investigator — 2nd department of dermatology and venereology,University of Athens, Greece; Ignatios Ikonomidis, MD,PhD, Principal Investigator — 2nd department of cardiology,University of Athens,Greece
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece